CLINICAL TRIAL: NCT04941326
Title: Investigation of the Effect of Spinal Mobilization and Respiration Techniques on Posture and Respiratory Function in Parkinson's Patients
Brief Title: The Effect of Spinal Mobilization on Respiratory Parameters in Parkinson's Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ramazan KURUL, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-ETB-001
Record Dates: First submitted 2021-06-15; First posted 2021-06-28 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease; Camptocormia; Restrictive Lung Disease
Keywords: Rehabilitation; Posture
MeSH Terms: conditions — Parkinson Disease; Camptocormia | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Two groups with sham control group
Who Masked: Participant, Outcomes Assessor
Masking Description: Participans and outcome assessors will be blinded to group allocation. Control group will receive same amount of sham mobilisations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal mobilization group (Active Comparator): Spinal mobilization will be applied to the application group for 4 weeks in addition to the treatments applied to the sham group
  Interventions: Other: Diaphragmatic stimulation treatment with PNF techniques; Other: Costal mobilization; Other: Breathing exercises; Other: Spinal mobilization
- Sham group (Sham Comparator): Diaphragmatic stimulation with proprioceptive neuromuscular facilitation techniques (PNF), diaphragmatic breathing techniques, costal mobilization treatments and sham mobilization will be applied to the sham group.
  Interventions: Other: Diaphragmatic stimulation treatment with PNF techniques; Other: Costal mobilization; Other: Breathing exercises; Other: Sham mobilization

INTERVENTIONS:
Other: Diaphragmatic stimulation treatment with PNF techniques — Thumbs and palms are placed along the cartilage edges of the lower ribs. At the end of the expiration, pressure and stretching are given as far into the chest and upwards as possible and a deep inspiration is requested immediately after the pressure. Both sides can be stimulated by repeated contraction technique. Hand holding positions may differ according to the patient's preference. If the patient's physical condition is not suitable, the application can be done with the thumbs, the thumb of the left hand for the right rib, and the thumb of the right hand for the left rib in the same lying position. The patient will be asked to do the application 2 times in a day with 10 repetitions for 4 weeks.
Other: Costal mobilization — In the supine position, the individual will place both hands around the 10-12th ribs and alternately apply an oblique push from the right and left sides to the opposite side. The exercise will be taught to the patient as training, and he will be asked to apply it 2 times a day with 20 repetitions for 4 weeks.
Other: Breathing exercises — It is done to increase the diaphragm activity of the individual and to suppress chest breathing. While lying in the supine position, the legs are placed in a hooked position, with one hand on the abdomen and the other on the chest, and the deep breath that is taken from the nose in 2 seconds is asked to exhale through the mouth in 4 seconds, while revealing as little movement in the chest as possible, the main movement is requested to be around the abdomen. The application will be given to the patient as a home program and he will be asked to do it 2 times a day with 5 repetitions for 4 weeks.
Other: Spinal mobilization — T12 vertebrae will be found by following the 12th rib in the prone position of the individual and spinous of L1 and L2 vertebrae will be determined with this reference. Then, small amplitude rotational movements in the vertebrae will be revealed by pushing in the anterior direction over the transverse processes. This application will be applied once a week for an average of 10 minutes for 4 weeks.
  Arms: Spinal mobilization group
Other: Sham mobilization — Sham pressures will be applied to the lumbar region of the patient, away from the vertebrae. This application will be applied once a week for an average of 10 minutes for 4 weeks.
  Arms: Sham group

SUMMARY:
Parkinson's patients suffer from respiratory distress for different reasons. It is thought that physiotherapy methods that have an indirect effect on the diaphragm can improve respiratory functions. The aim of this study is to investigate the effects of spinal mobilization and diaphragmatic breathing techniques on respiratory function.

DETAILED DESCRIPTION:
Respiratory complications are one of the most common causes of death in Parkinson's patients. Camptocormia may develop in Parkinson's disease and other pathological conditions involving the basal ganglia, which can be defined as an abnormal flexion of the thoracolumbar spine of 45° or more, which increases during walking or standing and disappears completely in the supine position. Parkinson's patients with camptocormia often complain of dyspnea, which can be attributed to reduced lung capacity due to limited chest expansion.

Restrictive changes due to respiratory muscle dysfunction in Parkinson's disease, upper airway obstruction, abnormal ventilatory control, and drug use such as levodopa have an effect on respiratory functions.

Restrictive dysfunction has been reported in 28-94% of patients with Parkinson's.

Postural disorders such as camptocormia can also lead to restriction. One study found that the lung volumes of Parkinson's disease patients with camptocormia decreased, although it was not associated with major clinical changes.

Diaphragmatic dyskinesia in Parkinson's patients may also lead to a restrictive deterioration in respiratory functions.

Studies examining the effects of chest and diaphragm mobilization on spirometric parameters in patients with cerebral palsy reported that the applied mobilization and soft tissue techniques improved FEV1 and FVC. The effect of indirect diaphragmatic treatments with vertebral mobilization in individuals with Parkinson's who are at risk of experiencing restrictive respiratory problems is unknown. The aim of this study is to examine the effects of spinal mobilization techniques for the diaphragm on respiratory function parameters and posture.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with Parkinson's disease
* Volunteering to participate in the study
* Modified Medical Research Council (MMRC) score >2

Exclusion Criteria:

* Those with COVID-19
* Diseases that increase intra-abdominal pressure
* Diseases affecting diaphragmatic motility
* Those who had a recent thoracic or abdominal operation
* Those who have a parenchymal, pleural or chest wall mass that will cause restriction on a recent chest X-ray or CT will not be included in the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Test | Four weeks
  Respiratory function tests will be performed on all individuals with the MIR SPIROLAB II brand pulmonary function test device. In each measurement, the maneuvers will be repeated at least 3 times and the best values will be recorded. Forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1) results from the test will be used to calculate the ratio of FEV1 to FVC (FEV1/FVC) will be recorded. The combined FEV1/FVC ratio will be used as primary outcome.

SECONDARY OUTCOMES:
Spinal Mouse Evaluation | Four weeks
  The Spinal Mouse is a computer-aided, non-invasive, easy-to-use electromagnetic handheld device designed to measure the curvature of the spine in various positions. Validity-reliability studies of the Spinal Mouse were conducted. Spinal posture assessment will be performed in the sagittal position. All spinous processes will be detected by palpation, starting from the spinous process of the seventh cervical vertebra to the spinous process of the third sacral vertebra by the physiotherapist. Measurements are planned to be performed in two different positions;
  * the individual is in a standing upright position.
  * the individual is asked to perform maximum body flexion
Camptocormia and Range of Motion Evaluations | Four weeks
  Postural deviations of the spine will be recorded through photographs taken from the side and back in the standing position. Flexion of the individual more than 45° from the thoracolumbar spine will be recorded as the presence of camptocormia.
  • Evaluation of the spine from a lateral view; The baseline is drawn perpendicular to the ground and passing behind the 5th lumbar spine. The body line is drawn to pass through the 1st thoracic vertebra and the 5th lumbar vertebra. The angle between the two lines is measured.
  The flexion angle and extension angle deficit of the knee joint will be measured with a goniometer.
Ultrasonography | Four weeks
  When the patient is in the supine position, by placing a transducer on the chest wall at the level of the right 9th intercostal space, diaphragmatic movement will be monitored during inspiration, and diaphragmatic thickness will be measured at the end of expiration and inspiration.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Kurul, Ph.D, Principal Investigator — Abant Izzet Baysal University
Locations (2):
- Turkey (Türkiye) (2):
  - Abant Izzet Baysal University Faculty of Health Science, Bolu
  - AIBU Physical Therapy and Rehabiltiation Department, Bolu

IPD SHARING:
Plan to Share IPD: No